CLINICAL TRIAL: NCT00002793
Title: PALLIATIVE LOCAL CHEMOTHERAPY FOR NON-RESECTABLE LIVER METASTASES FROM COLORECTAL CARCINOMA, A RANDOMISED PHASE III STUDY
Brief Title: Chemotherapy Via an Implantable Pump Compared With a Subcutaneous Port for Unresectable Liver Metastases in Patients With Resected Colorectal Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000064871; GER-ALM-03/95; EU-96007
Record Dates: First submitted 1999-11-01; First posted 2004-09-02 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2007-05

CONDITIONS: Colorectal Cancer; Metastatic Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer; liver metastases
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Colonic Neoplasms; Rectal Neoplasms | interventions — Fluorouracil; Leucovorin

INTERVENTIONS:
Drug: fluorouracil
Drug: leucovorin calcium

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug or giving the drugs in different ways may kill more tumor cells.

PURPOSE: Randomized phase III trial to compare the effectiveness of chemotherapy administered via an implantable pump with a subcutaneous port for unresectable liver metastases in patients with resected primary colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the efficacy of 2 schedules of fluorouracil/leucovorin given as a continuous intra-arterial infusion via an implantable pump vs. a subcutaneous port for unresectable liver metastases in patients with colorectal cancer. II. Compare the effect of each treatment on response rate, quality of life, and rate of technical complications in these patients.

OUTLINE: Randomized study. The following acronyms are used: CF Leucovorin calcium, NSC-3590 5-FU Fluorouracil, NSC-19893 Arm I: Single-Agent Chemotherapy with Drug Modulation. 5-FU; with CF. Weekly infusion via an implantable pump. Arm II: Single-Agent Chemotherapy with Drug Modulation. 5-FU; with CF. Weekly infusion via a subcutaneous infusion port. Arm III: Single-Agent Chemotherapy with Drug Modulation. 5-FU; with CF. Monthly infusion via an implantable pump. Arm IV: Single-Agent Chemotherapy with Drug Modulation. 5-FU; with CF. Monthly infusion via a subcutaneous infusion port.

PROJECTED ACCRUAL: A total of 336 patients will be entered in this multicenter study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Primary colorectal cancer with unresectable liver metastases Less than 75% involvement of the liver Radical resection of primary colon or rectal tumor required No local recurrence or extrahepatic metastases No portal vein thrombosis, ascites, or cirrhosis

PATIENT CHARACTERISTICS: Age: 18 to 76 Performance status: Karnofsky 70%-100% Hematopoietic: WBC greater than 3,000 Platelets greater than 100,000 Hepatic: Bilirubin no greater than 4 mg/dL Alkaline phosphatase no greater than 1,200 U/L Coagulation tests normal Renal: Creatinine no greater than 2.5 mg/dL Other: No prior malignancy

PRIOR CONCURRENT THERAPY: See Disease Characteristics No prior intra-arterial chemotherapy for liver metastases No prior hepatic chemoembolization At least 3 months since fluorouracil

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Estimated)
Dates: Start 1991-01

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Lorenz, MD, Study Chair — Johann Wolfgang Goethe University Hospital
Locations (1):
- Klinikum der J.W. Goethe Universitaet, Frankfurt, Germany